CLINICAL TRIAL: NCT07165327
Title: Injection Ports Versus Single-Use Needles for Insulin Administration in Diabetic Pregnancies: Impact on Dose Adherence and Patient Satisfaction
Brief Title: Injection Ports vs Single-Use Needles for Insulin in Pregnancy: Effects on Adherence and Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007824
Record Dates: First submitted 2025-08-20; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Gestatiaonl Diabetes Mellitus; Pregnancy; Diabetes in Pregnancy; Insulin Dependent Diabetes Mellitus; Insulin
Keywords: Gestational diabetes; Type 2 diabetes in pregnancy; Insulin administration; Injection port; Single-use needles; Dose adherence; Patient satisfaction; Insulin delivery devices; Pregnancy diabetes management
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 1; Insulin Resistance; Patient Satisfaction | interventions — Vascular Access Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Injection port (Experimental): Participants in this arm will administer all prescribed insulin doses using an injection port device for two weeks. The port will be inserted and replaced according to manufacturer instructions, typically every 3 days. Insulin will be delivered through the port using standard syringes or insulin pens, eliminating the need for multiple daily needle sticks. Participants will continue routine glucose monitoring as directed by their clinical care team.
  Interventions: Device: Injection Port for Insulin Administration
- Single-use insulin needles (Active Comparator): Participants in this arm will administer all prescribed insulin doses using standard single-use disposable needles for two weeks. Each injection will require a new sterile needle, consistent with routine clinical practice for insulin delivery in pregnancy. Participants will continue routine glucose monitoring as directed by their clinical care team.
  Interventions: Device: Single-Use Insulin Needles

INTERVENTIONS:
Device: Injection Port for Insulin Administration — For two weeks, participants will use an injection port device for all prescribed insulin doses during pregnancy. The port is inserted and replaced approximately every 3 days. Insulin is delivered through the port using standard syringes or insulin pens, eliminating the need for multiple daily needle sticks.
  Other Names: i-port; Insulin Port Device
  Arms: Injection port
Device: Single-Use Insulin Needles — For two weeks, participants will use standard single-use disposable needles for all prescribed insulin doses during pregnancy. A new sterile needle will be used for each injection, consistent with routine clinical practice.
  Other Names: Disposable Needles; Standard Insulin Needles
  Arms: Single-use insulin needles

SUMMARY:
This study wants to find out if using an injection port to give insulin during pregnancy helps people take their insulin more regularly and feel better about their care.

When someone has diabetes during pregnancy, it's very important to keep their blood sugar levels in a healthy range. This usually means checking blood sugar often and giving insulin through shots. But giving many shots each day can be hard and uncomfortable.

An injection port is a small device placed on the skin that lets patients give insulin through the same spot without poking themselves each time. This may make taking insulin easier and less painful.

Feeling comfortable with how insulin is given may help people stick to their treatment plan and have better health during pregnancy. Injection ports have already helped other patients, including pregnant people who needed other medications, but they haven't been studied for insulin use during pregnancy. This study will look at how pregnant patients with diabetes feel about using injection ports for insulin.

DETAILED DESCRIPTION:
Diabetes management during pregnancy is crucial for both maternal and fetal health, requiring frequent blood glucose monitoring and insulin administration. Traditional methods of insulin injection involve up to 5 insulin injections per day. These methods, while effective, can be burdensome, and many patients desire to avoid frequent injections.

Injection ports are small, single-use, prescription medical devices designed to simplify insulin or other subcutaneous medication delivery. They consist of a soft cannula that sits under the skin for up to 72 hours and a resealable septum through which multiple injections can be administered without repeated needle sticks. The I-port is an injection port that is FDA approved for use in the United States, but is rarely used in clinical practice, largely because it is not typically covered by insurance.

Given the importance of management of diabetes throughout pregnancy, patient satisfaction with insulin delivery methods may play a significant role in treatment adherence and overall health outcomes. The use of injection ports has been shown to improve patient satisfaction in pregnant patients requiring heparin administration in pregnancy, as well as improve patient experiences for insulin administration in non-pregnant populations. However, there are no studies that have evaluated the use of injection ports for insulin administration in pregnancy. This study aims to assess patient satisfaction with the use of injection ports for insulin administration among pregnant patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus or gestational diabetes who require a multi-dose insulin regimen

Exclusion Criteria:

* T1DM, primary language non-English or Spanish, use of an insulin pump

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Compliance with insulin administration | Two weeks
  Patients' compliance with their insulin administration during each arm will be assessed by determining the total number of insulin doses that were missed.
Patient satisfaction | Two weeks
  Patients' satisfaction with each method of insulin administration will be determined used the Insulin Delivery Satisfaction Survey

SECONDARY OUTCOMES:
Glucose control | Two weeks
  In each arm, patients' overall glucose control will be assessed by determining their percent time in range, mean fasting glucose (mg/dL), and mean postprandial glucose (mg/dL).
Hypoglycemia episodes | Two weeks
  Patients will be assessed on the frequency of hypoglycemia episodes in each arm
Adverse reactions | Two weeks
  Patients will be assessed for adverse reactions with each regimen, including allergic reactions or infections
Device malfunctions | Two weeks
  In each arm, patients will be asked if they experienced any device malfunctions and if so, what did they experience

CONTACTS AND LOCATIONS:
Overall Officials: Lorie Harper, Principal Investigator — University of Texas at Austin, Dell Medical School
Locations (1):
- University of Texas at Austin, Dell Medical School, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided